CLINICAL TRIAL: NCT02789137
Title: PROSPECTIVE, MULTICENTRE, OBSERVATIONAL STUDY ON FATIGUE- AND HAND-FOOT SYNDROME-RELATED QUALITY OF LIFE IN PATIENTS WITH METASTATIC RENAL CELL CARCINOMA RECEIVING A TYROSINE KINASE INHIBITOR AS FIRST-LINE TREATMENT (TROYA STUDY).
Brief Title: Study On Fatigue- And Hand-Foot Syndrome-Related Quality Of Life In Patients With Metastatic Renal Cell Carcinoma Receiving A Tyrosine Kinase Inhibitor as First-Line Treatment
Acronym: TROYA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181218; TROYA (Other: Alias Study Number)
Record Dates: First submitted 2016-05-17; First posted 2016-06-02 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: metastatic renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to know about the quality of life of patients with metastatic renal cell carcinoma who are being treated with sunitinib, pazopanib or sorafenib, and who suffer from fatigue and hand-foot syndrome, with personal inter-variability, and to explore measures that can be taken in terms of both everyday lifestyle and treatment to mitigate or cure such side effects that affect patients.

DETAILED DESCRIPTION:
Prospective, multicentre, observational study in patients with metastatic renal cell carcinoma (mRCC) receiving a tyrosine kinase inhibitor as first-line treatment according to routine clinical practice, designed to evaluate the incidence of fatigue and hand-foot syndrome in order to determine how these affect the baseline characteristics of the patient and his/her disease (age, gender, baseline status, tumour histology, etc.) and the patient's lifestyle as such side effects develop.

An exploratory analysis will be performed of measures that clinicians may adopt to improve patients' quality of life with regards to daytime naps, medication administration time, off-treatment periods, dose reductions and treatment breaks.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old and diagnosed with metastatic RCC who, in the investigator's opinion, are candidates for starting first-line treatment with a tyrosine kinase inhibitor according to routine clinical practice.
* Patients who have no contraindications to the treatment.
* Baseline ECOG ≤ 2.
* Patients who are able to give informed consent on their own without the need for a legal representative.
* Committed patients who are able to complete the quality of life questionnaires and patient diary on their own without the need for a legal representative.

Exclusion Criteria:

* Patients who are not candidates for first-line treatment with a tyrosine kinase inhibitor.
* Patients who are receiving the treatment as second-line or subsequent therapy.
* Untreated hypothyroidism.
* Untreated severe anaemia.
* Pregnancy or breast-feeding.
* Myocardial infarction or cerebrovascular accidents (CVA) within the last 6 months.
* Severe hepatic impairment.
* Concomitant use of potent inhibitors or inducers that interact with hepatic cytochrome CYP3A4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A population of 100 patients aged 18 years or over and diagnosed with metastatic renal cell carcinoma who are to start first-line treatment with a tyrosine kinase inhibitor according to routine clinical practice is to be studied
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- Spain (23):
  - Hospital Arquitecto Marcide de Ferrol, Ferrol, A Coruña
  - Hospital Asil de Granollers, Granollers, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Galdakano, Usansolo, Bizkaia
  - Complejo Hospitalario la Mancha Centro, Alcázar de San Juan, Ciudad REAL
  - Hospital Universitari Son Espases, Palma, Mallorca
  - Hospital Universitario Sant Joan de Reus / Servicio de Oncología Médica, Reus, Tarragona
  - H. Universitario Infanta Cristina, Badajoz
  - Hospital Vall de Hebrón, Barcelona
  - Hospital Universitario Ciudad Real, Ciudad Real
  - H. Reina Sofía de Cordoba, Córdoba
  - ICO Girona (Hospital Dr.Josep Trueta), Girona
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Hospitalario de León, León
  - Hospital Universitario La Princesa / Servicio de Oncología Médica, Madrid
  - Complejo Hospitalario Ourense. Hospital Santa María Nai, Ourense
  - Hospital General de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Canarias, Santa Cruz de Tenerife
  - Hospital de Sant Pau i Santa Tecla, Tarragona
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - H Clínico Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged above or equal to 18 years, who were diagnosed with metastatic renal cell carcinoma (mRCC), and were to initiate tyrosine kinase inhibitor (TKI) as first-line treatment as per normal routine healthcare practice in real world were included in this prospective, observational study. Participants were to be followed up for at least 9 months after treatment initiation and till they switched to second line treatment before end of the study (maximum duration of 3.8 years).
Groups:
- Tyrosine Kinase Inhibitor: Participants diagnosed with mRCC who received TKI as first line treatment, prescribed by physician, in real world practice were observed in this study.
Period: Overall Study
Arm/Group | Tyrosine Kinase Inhibitor
Started | 111
Completed | 53
Not Completed | 58
Not completed — Dropped out/Died | 58

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data was collected and analyzed in this study.
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Eastern Cooperative Oncology Group Performance Status (ECOG PS) Less Than or Equal to (<=) 2 [Count of Participants; unit: Participants] — ECOG PS: used to measure quality of life of oncology patients with scores running from 0 to 5; where 0= fully active, able to carry on all pre-disease performance without restriction; 1= restricted in physically strenuous activity, ambulatory, able to carry out light or sedentary work; 2= ambulatory, capable of all self-care, unable to carry out any work activity, up greater than (>)50 percent (%) of waking hours; 3= capable of only limited self-care, confined to bed or chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5= dead.
  Participants
    0 | 55
    1 | 45
    2 | 11
Heng Prognostic Criteria [Count of Participants; unit: Participants] — Heng prognostic model identified Karnofsky performance status (KPS) of less than (<) 80 at treatment initiation, period from mRCC diagnosis to previous systemic treatment <1 year, anemia, hypercalcemia, neutrophilia, thrombocythemia as independent poor prognostic factors. Participants classified into prognosis group: favorable(0 factor), intermediate(1-2 factors), poor(3-6 factors). KPS measured ability of participants with cancer to perform ordinary tasks. KPS scores range: 0 percent (%) (dead) to 100% (normal, no complaint). High score=participant better able to carry out daily activities.
  Participants
    Favourable | 28
    Intermediate | 57
    Poor prognosis | 26
Site of Metastasis [Count of Participants; unit: Participants] — Here, number of participants were classified according to type of metastatic sites.
  Participants
    Lung | 73
    Brain | 3
    Nodes | 38
    Bone | 29
    Liver | 26
    Kidney | 9
    Other | 32
Number of Metastatic Sites [Count of Participants; unit: Participants] — Here, number of participants were classified according to number of metastatic sites.
  Participants
    1 | 47
    2 | 36
    3 | 19
    4 | 6
    5 | 3
Histological Type [Count of Participants; unit: Participants] — Here, number of participants were classified according to type of histology as clear cell, non-clear cell (chromophobe, papillary type 1, papillary type 2), mixed, and sarcomatoid. Participants whose histology was not performed were reported as "not performed".
  Participants
    Clear cell | 86
    Chromophobe | 3
    Papillary type 1 | 4
    Papillary type 2 | 5
    Mixed | 3
    Sarcomatoid | 2
    Not performed | 8
Smoking Status [Count of Participants; unit: Participants] — Here, number of participants were classified according to smoking status as do not smoke, smoke, occasionally smoke and was a former smoker (did not smoke from less than [<] 6 months).
  Participants
    No | 79
    Yes | 20
    Occasional | 1
    Former Smoker | 11
Time Elapsed From the Time of Diagnosis of the Disease [Mean (Standard Deviation); unit: Months] — Here, the time elapsed since the moment of the initial diagnosis of the disease until the inclusion of the participant in the study was calculated as the difference between the disease diagnosis date and the baseline visit date.
  Months | 31.5 (56.9)
Time Elapsed From the Time of Advanced Diagnosis of the Disease [Mean (Standard Deviation); unit: Months] — Here, the time elapsed since the moment of the diagnosis of the advanced disease until the inclusion of the participant in the study was calculated as the difference between the date of the advanced stage diagnosis and the baseline visit date.
  Months | 2.6 (4.8)
Number of Participants Categorized According to Tyrosine Kinase Inhibitor Dose and Treatment Regimen [Count of Participants; unit: Participants] — Here, number of participants were classified according to type of TKI with dose specification and the treatment regimen received as the first line treatment. "2/1" regimen meant 14 days on drug and 7 days without drug. "4/2" regimen meant 28 days on drug and 14 days without drug.
  Participants
    Pazopanib 800 mg daily without rest days | 11
    Sunitinib 50 mg, Regimen 4/2 | 83
    Sunitinib 50 mg, Regimen 2/1 | 10
    Sunitinib 37.5 mg, Regimen 4/2 | 2
    Sunitinib 37.5 mg, Regimen 2/1 | 3
    Sunitinib 25 mg, Regimen 2/1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized According to the Napping Habits for All Participants at Baseline
Description: In this outcome measure, number of participants were classified according to their habit of taking daytime rest (naps) as never, always and sometimes. Never is defined as someone who does not take any daytime nap, always is defined as someone who takes daytime naps daily and sometimes is defined as someone who takes daytime naps on weekends or on holidays.
Time Frame: Baseline
Population: Analysis population included all eligible participants who were included in this study. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 86
Participants
  Never | 22
  Always | 33
  Sometimes | 31

2. Primary Outcome: Number of Participants Categorized According to the Napping Habits for All Participants at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 63
Participants
  Never | 18
  Always | 24
  Sometimes | 21

3. Primary Outcome: Number of Participants Categorized According to the Napping Habits for All Participants at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 45
Participants
  Never | 18
  Always | 15
  Sometimes | 12

4. Primary Outcome: Number of Participants Categorized According to the Napping Habits for All Participants at Week 36
Description: as for outcome 1
Time Frame: Week 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 41
Participants
  Never | 16
  Always | 16
  Sometimes | 9

5. Primary Outcome: Number of Participants Categorized According to Association Between the Practice of Aerobic Physical Exercise and Fatigue at Baseline
Description: In this outcome measure, number of participants were classified according to the presence or absence of fatigue based on their habit of performing aerobic physical exercise as never, always and sometimes.
Time Frame: Baseline
Population: Analysis population included all eligible participants who were included in this study. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 87
Participants
  Fatigue: Yes: number analyzed (Participants) | 17
  Fatigue: Yes: Never Exercise | 10
  Fatigue: Yes: Always Exercise | 0
  Fatigue: Yes: Sometimes Exercise | 7
  Fatigue: No: number analyzed (Participants) | 70
  Fatigue: No: Never Exercise | 34
  Fatigue: No: Always Exercise | 14
  Fatigue: No: Sometimes Exercise | 22

6. Primary Outcome: Number of Participants Categorized According to Association Between the Practice of Aerobic Physical Exercise and Fatigue at Week 12
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 62
Participants
  Fatigue: Yes: number analyzed (Participants) | 30
  Fatigue: Yes: Never Exercise | 14
  Fatigue: Yes: Always Exercise | 6
  Fatigue: Yes: Sometimes Exercise | 10
  Fatigue: No: number analyzed (Participants) | 32
  Fatigue: No: Never Exercise | 9
  Fatigue: No: Always Exercise | 12
  Fatigue: No: Sometimes Exercise | 11

7. Primary Outcome: Number of Participants Categorized According to Association Between the Practice of Aerobic Physical Exercise and Fatigue at Week 24
Description: as for outcome 5
Time Frame: Week 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 47
Participants
  Fatigue: Yes: number analyzed (Participants) | 25
  Fatigue: Yes: Never Exercise | 13
  Fatigue: Yes: Always Exercise | 5
  Fatigue: Yes: Sometimes Exercise | 7
  Fatigue: No: number analyzed (Participants) | 22
  Fatigue: No: Never Exercise | 10
  Fatigue: No: Always Exercise | 5
  Fatigue: No: Sometimes Exercise | 7

8. Primary Outcome: Number of Participants Categorized According to Association Between the Practice of Aerobic Physical Exercise and Fatigue at Week 36
Description: as for outcome 5
Time Frame: Week 36
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 41
Participants
  Fatigue: Yes: number analyzed (Participants) | 8
  Fatigue: Yes: Never Exercise | 4
  Fatigue: Yes: Always Exercise | 1
  Fatigue: Yes: Sometimes Exercise | 3
  Fatigue: No: number analyzed (Participants) | 33
  Fatigue: No: Never Exercise | 19
  Fatigue: No: Always Exercise | 5
  Fatigue: No: Sometimes Exercise | 9

9. Primary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Baseline
Description: FACIT-F was a 13-item questionnaire which assessed self-reported fatigue and its impact upon daily activities and function. Participants responded to each item on a 5-point scale based on their experience of fatigue during the past 7 days (0= not at all; 1= a little bit; 2= somewhat; 3= quite a bit; 4= very much). FACIT-F score was calculated by summing the 13 items (range 0 [not at all] to 52 [very much]); higher scores represented less fatigue and better status of participants.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 86
Units on a scale | 40.0 (9.6)

10. Primary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 6
Description: as for outcome 9
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 83
Units on a scale | 34.7 (11.4)

11. Primary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 12
Description: as for outcome 9
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 61
Units on a scale | 36.4 (10.6)

12. Primary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 18
Description: as for outcome 9
Time Frame: Week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 57
Units on a scale | 35.3 (11.5)

13. Primary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 24
Description: as for outcome 9
Time Frame: Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 43
Units on a scale | 36.3 (11.1)

14. Primary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 30
Description: as for outcome 9
Time Frame: Week 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 43
Units on a scale | 34.9 (11.3)

15. Primary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 36
Description: as for outcome 9
Time Frame: Week 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 43
Units on a scale | 35.5 (10.2)

16. Primary Outcome: Number of Participants Classified According to Time of Taking Treatment at Week 1
Description: In this outcome measure, the number of participants were classified on the basis of the time of taking the oral medication - "morning, afternoon or night". Morning was anytime between 7 am to 12 pm. Afternoon was anytime between 1 pm and 7 pm. Night was anytime between 8 pm to 6 am. Participants who did not take medication were also classified.
Time Frame: Week 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 86
Participants
  Morning | 39
  Afternoon | 31
  Night | 15
  Participant did not take medication in this week | 1

17. Primary Outcome: Number of Participants Classified According to Time of Taking Treatment at Week 6
Description: as for outcome 16
Time Frame: Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 82
Participants
  Morning | 19
  Afternoon | 13
  Night | 7
  Participant did not take medication in this week | 43

18. Primary Outcome: Number of Participants Classified According to Time of Taking Treatment at Week 12
Description: as for outcome 16
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 63
Participants
  Morning | 21
  Afternoon | 10
  Night | 10
  Participant did not take medication in this week | 22

19. Primary Outcome: Number of Participants Classified According to Time of Taking Treatment at Week 18
Description: as for outcome 16
Time Frame: Week 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 58
Participants
  Morning | 19
  Afternoon | 9
  Night | 6
  Participant did not take medication in this week | 24

20. Primary Outcome: Number of Participants Classified According to Time of Taking Treatment at Week 24
Description: as for outcome 16
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 45
Participants
  Morning | 12
  Afternoon | 8
  Night | 12
  Participant did not take medication in this week | 13

21. Primary Outcome: Number of Participants Classified According to Time of Taking Treatment at Week 30
Description: as for outcome 16
Time Frame: Week 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 45
Participants
  Morning | 12
  Afternoon | 9
  Night | 10
  Participant did not take medication in this week | 14

22. Primary Outcome: Number of Participants Classified According to Time of Taking Treatment at Week 36
Description: as for outcome 16
Time Frame: Week 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 41
Participants
  Morning | 10
  Afternoon | 8
  Night | 7
  Participant did not take medication in this week | 16

23. Primary Outcome: Number of Participants Categorized According to Number of Changes to Dose Per Treatment Cycle During 9 Months of Follow-up
Description: In this outcome measure, number of participants were classified according to the number of changes to dose that is (i.e). 0, 1 or 2 occurred per treatment cycle during 9 months of follow-up.
Time Frame: During 9 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 101
Participants
  Changes to Dose Occurred in Cycle 1: 0 | 82
  Changes to Dose Occurred in Cycle 1: 1 | 19
  Changes to Dose Occurred in Cycle 1: 2 | 0
  Changes to Dose Occurred in Cycle 2: number analyzed (Participants) | 94
  Changes to Dose Occurred in Cycle 2: 0 | 69
  Changes to Dose Occurred in Cycle 2: 1 | 25
  Changes to Dose Occurred in Cycle 2: 2 | 0
  Changes to Dose Occurred in Cycle 3: number analyzed (Participants) | 72
  Changes to Dose Occurred in Cycle 3: 0 | 55
  Changes to Dose Occurred in Cycle 3: 1 | 17
  Changes to Dose Occurred in Cycle 3: 2 | 0
  Changes to Dose Occurred in Cycle 4: number analyzed (Participants) | 68
  Changes to Dose Occurred in Cycle 4: 0 | 60
  Changes to Dose Occurred in Cycle 4: 1 | 7
  Changes to Dose Occurred in Cycle 4: 2 | 1
  Changes to Dose Occurred in Cycle 5: number analyzed (Participants) | 55
  Changes to Dose Occurred in Cycle 5: 0 | 46
  Changes to Dose Occurred in Cycle 5: 1 | 9
  Changes to Dose Occurred in Cycle 5: 2 | 0
  Changes to Dose Occurred in Cycle 6: number analyzed (Participants) | 53
  Changes to Dose Occurred in Cycle 6: 0 | 49
  Changes to Dose Occurred in Cycle 6: 1 | 4
  Changes to Dose Occurred in Cycle 6: 2 | 0

24. Primary Outcome: Number of Participants Categorized According to Number of Interruptions to Dose Occurred in Each Treatment Cycle During 9 Months of Follow-up
Description: In this outcome measure, number of participants were classified according to the number of interruptions to dose i.e. 0, 1, 2, 3 or 4 occurred in each treatment cycle during 9 months follow-up.
Time Frame: During 9 months
Population: Analysis population included all eligible participants who were included in this study. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 111
Participants
  Interruptions in Cycle 1: number analyzed (Participants) | 101
  Interruptions in Cycle 1: 0 | 76
  Interruptions in Cycle 1: 1 | 25
  Interruptions in Cycle 1: 2 | 0
  Interruptions in Cycle 1: 3 | 0
  Interruptions in Cycle 1: 4 | 0
  Interruptions in Cycle 2: number analyzed (Participants) | 94
  Interruptions in Cycle 2: 0 | 73
  Interruptions in Cycle 2: 1 | 16
  Interruptions in Cycle 2: 2 | 5
  Interruptions in Cycle 2: 3 | 0
  Interruptions in Cycle 2: 4 | 0
  Interruptions in Cycle 3: number analyzed (Participants) | 71
  Interruptions in Cycle 3: 0 | 59
  Interruptions in Cycle 3: 1 | 9
  Interruptions in Cycle 3: 2 | 3
  Interruptions in Cycle 3: 3 | 0
  Interruptions in Cycle 3: 4 | 0
  Interruptions in Cycle 4: number analyzed (Participants) | 67
  Interruptions in Cycle 4: 0 | 58
  Interruptions in Cycle 4: 1 | 7
  Interruptions in Cycle 4: 2 | 2
  Interruptions in Cycle 4: 3 | 0
  Interruptions in Cycle 4: 4 | 0
  Interruptions in Cycle 5: number analyzed (Participants) | 54
  Interruptions in Cycle 5: 0 | 39
  Interruptions in Cycle 5: 1 | 12
  Interruptions in Cycle 5: 2 | 2
  Interruptions in Cycle 5: 3 | 1
  Interruptions in Cycle 5: 4 | 0
  Interruptions in Cycle 6: number analyzed (Participants) | 52
  Interruptions in Cycle 6: 0 | 41
  Interruptions in Cycle 6: 1 | 10
  Interruptions in Cycle 6: 2 | 1
  Interruptions in Cycle 6: 3 | 0
  Interruptions in Cycle 6: 4 | 0

25. Primary Outcome: Number of Participants With Best Response Per Response Evaluation Criteria for Solid Tumours Version 1.1. (RECIST v1.1)
Description: Best response was recorded from start of treatment with TKI until best complete response (CR), partial response (PR), stable disease (SD) or disease progression (DP) was achieved. RECIST v1.1, a) CR: disappearance of all lesions; any pathological lymph nodes (target lesions [TLs]) or non-target lesions (non-TLs) must have reduction in short axis to <10 mm; normalization of tumor marker level for non-TLs; b) PR: >=30% decrease in sum of diameter of all TLs, taking as reference baseline sum of diameters; c) DP: >=20% increase in sum of diameter of all TLs, taking as reference the smallest sum on study (including baseline measurement), sum must also be absolute increase of >=5 mm. Unequivocal progression of existing non TLs. Appearance of at least 1 new lesion; d) SD: neither sufficient shrinkage to qualify for PR nor sufficient increase in lesions to qualify for PD referring smallest sum diameter. Participant whose best response was not determined were classified as "Undetermined".
Time Frame: From start of treatment with TKI until first documented best response of CR, PR, SD or DP (approximately maximum up to 3.8 years)
Population: Analysis population included all eligible participants who were included in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 111
Participants
  CR | 0
  PR | 42
  SD | 29
  DP | 28
  Undetermined | 12

26. Primary Outcome: Mean Duration of Treatment
Description: In this outcome measure, the mean duration of treatment was calculated and reported below.
Time Frame: From start of treatment till end of treatment (approximately maximum up to 3.8 years)
Population: Analysis population included all eligible participants who were included in this study.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 111
Months | 8.9 (7.7)

27. Primary Outcome: Time to Treatment Failure (TTF) After Initiation of Tyrosine Kinase Inhibitor Therapy
Description: TTF was defined as the time from the start of treatment with a TKI to tumour progression, treatment discontinuation for any reason or death from any cause. Participants who did not had the event were censored on the date of their final follow-up. Per RECIST 1.1, tumour progression: >=20% increase in sum of diameter of all measured target lesions, taking as reference smallest sum on study (including baseline measurement) of diameter of all target lesions, sum must also demonstrate an absolute increase of >=5 mm. Unequivocal progression of existing non target lesions. Appearance of at least 1 new lesion.
Time Frame: From start of treatment with a TKI to tumour progression, treatment discontinuation for any reason or death from any cause or till follow-up in case of no event (approximately maximum up to 3.8 years)
Population: Analysis population included all eligible participants who were included in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 111
Months | 6.9 [4.6 to 9.2]

28. Primary Outcome: Number of Participants Categorized According to Number of Treatment Cycles Received
Description: In this outcome measure, number of participants were classified according to number of treatment cycles received.
Time Frame: From start of treatment till end of treatment (approximately maximum up to 3.8 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 88
Participants
  0 cycles | 2
  1 cycle | 10
  2 cycles | 21
  3 cycles | 8
  4 cycles | 12
  5 cycles | 3
  6 cycles | 4
  7 cycles | 9
  8 cycles | 5
  9 cycles | 1
  10 cycles | 4
  11 cycles | 1
  12 cycles | 1
  13 cycles | 1
  14 cycles | 2
  15 cycles | 1
  17 cycles | 1
  19 cycles | 1
  25 cycles | 1

29. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the start of treatment with a TKI to tumour progression or death for any reason. Participants who, did not had the event were censored on the date of their final follow-up. Per RECIST v1.1, tumour progression: >=20% increase in sum of diameter of all measured target lesions, taking as reference smallest sum on study (including baseline measurement) of diameter of all target lesions, sum must also demonstrate an absolute increase of >=5 mm. Unequivocal progression of existing non target lesions. Appearance of at least 1 new lesion.
Time Frame: From start of treatment with a TKI to tumour progression or death for any reason or till follow-up in case of no event (approximately maximum up to 3.8 years)
Population: Analysis population included all eligible participants who were included in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 111
Months | 9.3 [6.2 to 10.9]

30. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved CR or PR. Per RECIST V1.1, a) CR: disappearance of all lesions; any pathological lymph nodes (target lesions or non-target lesions) must have reduction in short axis to <10 mm; normalization of tumor marker level for non-TLs; b) PR: >=30% decrease in sum of diameter of all target lesions, taking as reference baseline sum of diameters.
Time Frame: From start of treatment with TKI until first documented CR or PR (approximately maximum up to 3.8 years)
Population: Analysis population included all eligible participants who were included in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 111
Percentage of participants | 37.8

31. Primary Outcome: Duration of Response (DOR)
Description: In participants who achieved CR or PR, DOR was defined as the duration from the documentation date of CR or PR to the first day when DP was observed. Per RECIST V1.1, a) CR: disappearance of all lesions; any pathological lymph nodes (target lesions or non-target lesions must have reduction in short axis to <10 mm; normalization of tumor marker level for non-target lesions; b) PR: >=30% decrease in sum of diameter of all target lesions, taking as reference baseline sum of diameters; c) DP: >=20% increase in sum of diameter of all measured target lesions, taking as reference smallest sum on study (including baseline measurement), sum must also demonstrate an absolute increase of >=5 mm. Unequivocal progression of existing non TLs. Appearance of at least 1 new lesion.
Time Frame: From day of documented CR or PR to the first day that DP was observed (approximately maximum up to 3.8 years)
Population: Analysis population included all eligible participants who were included in this study. Here 'Overall Number of Participants Analyzed' signifies participants with documented CR or PR.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 42
Months | 11.8 (7.3)

32. Primary Outcome: Number of Participants With Fatigue Event Graded Per Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per CTCAE version 4, Grade 1= mild AE; Grade 2= moderate AE; Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE. In this outcome measure number of participants with fatigue event were classified into following: CTCAE grade 1 to 2 and CTCAE grade 3 to 4.
Time Frame: During 9 months
Population: Analysis population included all eligible participants who were included in this study. Here, "Overall Number of Participants Analyzed" signifies participants with fatigue event.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 6
Participants
  Grade 1-2 | 6
  Grade 3-4 | 0

33. Primary Outcome: Number of Participants With Hand Foot Syndrome Event Graded Per Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per CTCAE version 4, Grade 1= mild AE; Grade 2= moderate AE; Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE. In this outcome measure number of participants with hand foot syndrome event were classified into following: CTCAE grade 1 to 2 and CTCAE grade 3 to 4.
Time Frame: During 9 months
Population: Analysis population included all eligible participants who were included in this study. Here, "Overall Number of Participants Analyzed" signifies participants with hand foot syndrome event.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 32
Participants
  Grade 1-2 | 30
  Grade 3-4 | 2

34. Primary Outcome: Number of Participants With Palmar-Plantar Erythrodysaesthesia (HFS) Event Graded Per CTCAE Version 4.0 at Week 12
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per CTCAE version 4, Grade 1= mild AE; Grade 2= moderate AE; Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE. In this outcome measure number of participants with HFS event graded per CTCAE version 4.0 at Week 12 are reported.
Time Frame: Week 12
Population: Analysis population included all eligible participants who were included in this study. Here, 'Overall Number of Participants Analyzed' signifies participants with HFS event at Week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 19
Participants
  Grade 1 | 11
  Grade 2 | 7
  Grade 3 | 1

35. Primary Outcome: Number of Participants With Palmar-Plantar Erythrodysaesthesia (HFS) Event Graded Per CTCAE Version 4.0 at Week 24
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per CTCAE version 4, Grade 1= mild AE; Grade 2= moderate AE; Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE. In this outcome measure number of participants with HFS event graded per CTCAE version 4.0 at Week 24 are reported.
Time Frame: Week 24
Population: Analysis population included all eligible participants who were included in this study. Here, 'Overall Number of Participants Analyzed' signifies participants with HFS event at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 14
Participants
  Grade 1 | 11
  Grade 2 | 2
  Grade 3 | 1

36. Primary Outcome: Number of Participants With Palmar-Plantar Erythrodysaesthesia (HFS) Event Graded Per CTCAE Version 4.0 at Week 36
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per CTCAE version 4, Grade 1= mild AE; Grade 2= moderate AE; Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE. In this outcome measure number of participants with HFS event graded per CTCAE version 4.0 at Week 36 are reported.
Time Frame: Week 36
Population: Analysis population included all eligible participants who were included in this study. Here, 'Overall Number of Participants Analyzed' signifies participants with HFS event at Week 36.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor
Number analyzed (Participants) | 10
Participants
  Grade 1 | 8
  Grade 2 | 1
  Grade 3 | 1

ADVERSE EVENTS:
Time Frame: From start of treatment till end of treatment (approximately maximum up to 3.8 years)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Analysis population included all eligible participants whose data was collected and analyzed in this study.
Groups:
- Sunitinib: Participants diagnosed with mRCC who received either 4/2 regimen or 2/1 regimen of 50 mg or 37.5 mg or 25 mg dose of Sunitinib as first line treatment, prescribed by physician, in real world practice were observed in this study. "2/1" regimen meant 14 days on drug and 7 days without drug. "4/2" regimen meant 28 days on drug and 14 days without drug.
- Pazopanib: Participants diagnosed with mRCC who received 800 mg of Pazopanib per 24 hours continuously as first line treatment, prescribed by physician, in real world practice were observed in this study.
Arm/Group | Sunitinib | Pazopanib
All-Cause Mortality (participants affected / at risk) | 17/100 | 1/11
Serious Adverse Events (participants affected / at risk) | 23/100 | 5/11
Other Adverse Events (participants affected / at risk) | 82/100 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=100) | Pazopanib (N=11)
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Cardiotoxicity (Cardiac disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Oral mucosal disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Mucosal inflammation (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=100) | Pazopanib (N=11)
Anaemia (Blood and lymphatic system disorders) | 6 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 10 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 0
Hypothyroidism (Endocrine disorders) | 7 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 35 | 3
Dyspepsia (Gastrointestinal disorders) | 9 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Odynophagia (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral mucosal disorder (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Asthenia (General disorders) | 53 | 4
Fatigue (General disorders) | 5 | 1
Mucosal dryness (General disorders) | 3 | 0
Mucosal inflammation (General disorders) | 40 | 1
Oedema (General disorders) | 6 | 0
Pyrexia (General disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Ageusia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 16 | 1
Headache (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 3 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 28 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 18 | 0
Hypertension (Vascular disorders) | 21 | 1
Cardiotoxicity (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT02789137/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT02789137/SAP_001.pdf